CLINICAL TRIAL: NCT03417024
Title: Automated Breast Ultrasound Case Collection Registry
Status: Terminated | Type: Observational
Why Stopped: Change in business strategy
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 110.01-2016-GES-0001
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Subjects: All subjects will undergo scanning with both Automated Breast Ultrasound and Digital Breast Tomosynthesis devices.
  Interventions: Device: Automated Breast Ultrasound; Device: Digital Breast Tomosynthesis

INTERVENTIONS:
Device: Automated Breast Ultrasound — The ABUS system is designed to methodically scan a breast and capture multiple ultrasound images that can be rendered and reviewed in three dimensions.
Device: Digital Breast Tomosynthesis — Digital Breast Tomosynthesis (DBT) systems are designed to collect 3-dimensional x-ray images of breast tissues.

SUMMARY:
The contribution of automated breast ultrasound (ABUS) to the screening pathway for breast cancer is not fully understood. This prospective study aims to collect longitudinal data in women with dense breasts undergoing ABUS as a supplement to digital breast tomosynthesis (DBT). The data are intended for use in future research on the value and effectiveness of ABUS in routine clinical care.

Data will be collected from eligible women who have been prescribed or have completed DBT and ABUS, screening within a 30-day window. Radiologist evaluations and, when performed, outcomes of biopsy and/or laboratory testing will be recorded. Subjects will be followed for breast cancer status and results of any diagnostic breast exams and/or treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Are asymptomatic adult women (aged 18 years or older);
2. Are eligible to complete or have completed (within 30 days) screening ABUS and DBT exams per the site standard of care;1
3. Have heterogeneously dense and extremely dense breasts (BI-RADS C or D, respectively) or are determined to have dense breasts prior to the study on initial screening mammography;
4. Are able and willing to participate.

Exclusion Criteria:

1. Have a breast cancer diagnosis (with or without metastasis) or are being treated for breast cancer within the year prior to the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult women with dense breasts clinically referred for breast cancer screening.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Subjects
Started | 13
Completed | 0
Not Completed | 13
Not completed — Study Termination prior to follow-up | 11
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 5
  Race: Black, African American, or Negro | 7
  Race: Hispanic, Latino, or Spanish Origin | 1
  Race: Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Complete Breast Imaging Datasets
Time Frame: Up to 6 Years
Population: Study terminated prior to follow-up of any participants. No completed datasets were collected.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

2. Secondary Outcome: Type of Exams Performed Per Patient
Time Frame: Up to 6 years
Population: All exams performed for enrolled subjects
Measure: Number; unit: Exams completed
Arm/Group | All Subjects
Number analyzed (Participants) | 13
Exams completed
  ABUS | 11
  DBT | 12

3. Secondary Outcome: Breast Cancer Status
Time Frame: Up to 6 years
Population: 11 after withdrawals
Measure: Number; unit: Subjects with findings
Arm/Group | All Subjects
Number analyzed (Participants) | 11
Subjects with findings
  Initial Diagnosis (Cancer) | 0
  Initial Diagnosis (Non-Cancer) | 4

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT03417024/Prot_000.pdf